CLINICAL TRIAL: NCT01599559
Title: IELSG37: A Randomized, Open-label, Multicentre, Two-arm Phase III Comparative Study Assessing the Role of Involved Mediastinal Radiotherapy After Rituximab Containing Chemotherapy Regimens to Patients With Newly Diagnosed Primary Mediastinal Large B-Cell Lymphoma (PMLBCL)
Brief Title: Randomized, Open-label, Two-arms, Phase III Comparative Study Assessing the Role of Involved Mediastinal Radiotherapy After Rituximab Containing Chemotherapy Regimens to Patients With Newly Diagnosed Primary Mediastinal Large B-Cell Lymphoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IELSG37
Record Dates: First submitted 2012-05-10; First posted 2012-05-16 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Primary Mediastinal B-cell Lymphoma
Keywords: previously; untreated
MeSH Terms: interventions — Observation; Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- observation (Experimental): Follow up visits are scheduled from randomization. Patients will be seen at 3-months intervals for 24 months, then every 6 months until 5 years from randomization.
  Interventions: Other: observation
- mediastinal irradiation (Active Comparator): Radiotherapy will be delivered in this phase III protocol, as alternative to observation, as consolidation treatment in patients achieving a CR status (PET/CT scan negative) at the end of R-chemotherapy, with a total dose of 30 Gy.
  Interventions: Radiation: 3D-Conformal Radiotherapy (3D-CRT)

INTERVENTIONS:
Other: observation — observation
  Arms: observation
Radiation: 3D-Conformal Radiotherapy (3D-CRT) — Radiation treatment should start within 6-8 weeks after the end of chemotherapy.
  Arms: mediastinal irradiation

SUMMARY:
Primary mediastinal large B cell lymphoma is treated with a combination of chemotherapy and the monoclonal antibody rituximab (chemoimmunotherapy).

Following chemoimmunotherapy patients receive radiation therapy if they have residues which may be active tumour. However at the end of chemoimmunotherapy the majority of patients show tissue scarring that is not necessarily active tumor. In recent years, PET/CT has proved to be a good tool to accurately identify active tumor from scar tissue in patients treated for mediastinal lymphoma.The purpose of this trial is to test whether radiation therapy is really necessary in patients where PET/CT has shown that the tumor is no longer active. Therefore we will compare radiation treatment with careful observation.

Patients that at the end of conventional treatment of chemoimmunotherapy have a negative PET/CT (i.e., without residues suspected to contain active tumor), will randomly assigned to two different treatment groups: one treatment group will receive the radiation treatment, and the other treatment group will receive careful observation.

The trial is planned according to a non-inferiority design aimed at demonstrating that progression free survival after the experimental treatment (observation) is not worse than after the standard comparator (mediastinal irradiation.Participation in this study could spare patients with complete remission at the end of chemo immunotherapy (PET/CT negative) radiation therapy that may be unnecessary.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated primary mediastinal diffuse large B-cell lymphoma, CD20 positive.
* Patients must have histological confirmation of the diagnosis (it is recommended that the immunohistochemical panel includes: CD45, CD20, CD30, CD15, CD10, BCL6, BCL2, MUM-1), and in addition have a dominant mass within the anterior mediastinum.
* No evidence of extranodal disease outside the chest including spleen and bone marrow.
* Age at least 18 years.
* Fit to receive chemotherapy and radiotherapy with curative intent.
* Patients will be eligible if the treatment phase consisting in a Rituximab combined with any anthracycline-containing chemotherapy regimen without consolidation with autologous stem cell support (e.g., 6 cycles of CHOP14-21, DA-EPOCH, Mega-CHOP or 12 weeks of VACOP-B or MACOP-B).
* At least 6 courses of Rituximab should be administered
* Able and willing to give informed consent, and to undergo staging including PET scanning
* Willingness to comply with an appropriate contraceptive method in women of childbearing potential or men.
* Histological diagnostic material available for review.

Exclusion Criteria:

* History of malignancy other than squamous cell carcinoma, basal cell carcinoma of the skin or carcinoma in situ of the cervix within the last 5 years.
* Evidence of clinically significant cardiac disease at diagnosis, as defined by history of symptomatic ventricular arrhythmias, congestive heart failure or myocardial infarction within 12 months before study entry. Cardiac impairment due to local extension of lymphoma will not be an exclusion criterion in the absence of other cardiac disease.
* Known HIV-positive serology.
* Pregnant or lactating women.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2012-10 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2029-12-17 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 30 months from the randomization
  The primary outcome endpoint will be Progression Free Survival (PFS) in patients PET-negative after R-chemotherapy.
  Failure events for PFS are progression (defined as an increase in size of existing masses or the development of new sites of disease using the same radiological investigations CT or PET/CT and/or MRI - as for the pre-chemotherapy assessment) or death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years from registration
  OS is defined as the time from registration until death as a result of any cause until five years from registration
Long term toxicity | 10 years from registration
  Reporting of any adverse event which is judged in the opinion of investigator to be possibly treatment-related up to 10 years from randomization (including all cardiac and pulmonary events, relapses and second cancers and deaths)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Martelli, MD, Study Chair — Università La Sapienza (Rome - Italy); Andrew J Davies, MD, Study Chair — University of Southampton (UK); Mary Gospodarowicz, MD, Study Chair — Princess Margaret Hospital Toronto (Canada); Sally F Barrington, MD, Study Chair — St. Thomas' - London (UK); Alberto Biggi, MD, Study Chair — AO S. Croce e Carle, Cuneo (Italia); Annibale Versari, MD, Study Chair — S.Maria Nuova Hospital, Reggio Emilia (Italia); Gianni Ciccone, MD, Study Chair — CPO Torino (Italy); Stèphane Chauvie, MD, Study Chair — AO S. Crtoce e Carle - Cuneo (Italy); Luca Ceriani, MD, Study Chair — IOSI - Bellinzona (Switzerland)
Locations (85):
- United States (3):
  - Norton Cancer Institute, Louisville, Kentucky
  - Mayo Clinil Rocheser, Rochester, Minnesota
  - MD Anderson Cancer Center, Houston, Texas
- Centro de Hematologia y Oncologia Pavlovsky, Buenos Aires, Argentina
- Princess Margaret Hospital, Toronto, Canada
- Ruijin Hospital, Shanghai, China
- Czechia (4):
  - Faculty Hospital Brno, Brno
  - University Hospital, Hradec Králové
  - Faculty Hospital Kralovske Vinohrady, Prague
  - General University Hospital, Prague
- University of Duisburg-Essen, Campus Essen, Essen, Germany
- Italy (52):
  - A.O. SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Clinica di Ematologia Ospedali Riuniti "Umberto I", Ancona
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - A.O.U Policlinico Consorziale di Bari, Bari
  - Bari IRCCS Istituto Tumori, Bari
  - Ospedale Mons. Dimiccoli, Barletta
  - Ospedale Papa Giovanni Xxiii, Bergamo
  - Sant'Orsola Malpighi, Bologna
  - Comprensorio Sanitario di Bolzano, Bolzano
  - Spedali Civili, Brescia
  - Asl Uoc Ematologia A Perrino, Brindisi
  - Ospedale Businco, Cagliari
  - AO Garibaldi Nesima Catalia, Catania
  - Ospedale S. Croce e Carle, Cuneo
  - Unità Funzionale di Ematologia AOU Careggi, Florence
  - U.O. Ematologia Vito Fazzi, Lecce
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - SC Ematologia Azienda Ospedali Riuniti Papardo Piemonte, Messina
  - Istituto Scientifico San Raffaele, Milan
  - Milano Ieo, Milan
  - SC Ematologia AO Niguarda, Milan
  - AOU Policlinico di Modena, Modena
  - Ematologia Università degli Studi di Federico II, Napoli
  - Ospedale Umberto I, Nocera Inferiore
  - Azienda Ospedaliera Universitaria, Padua
  - Ospedali Riuniti Villa Sofia, Palermo
  - AOU di Parma, Parma
  - Fondazione IRCCS S. Matteo, Pavia
  - S.C. Ematologia Ospedale S. Marid Della Misericordia, Perugia
  - Ospedale Civile di Pescara, Pescara
  - Ospedale Civico Guglielmo di Saliceto, Piacenza
  - Ospedale San Carlo di Potenza, Potenza
  - U.O. Oncologia Ematologia Ospedale S. Maria Delle Croci, Ravenna
  - A.O. Bianchi-Melacrino-Morelli, Divisione di Ematologia, Reggio Calabria
  - ICCRS Azienda Ospedaliera Arcipedale "Santa Maria Nuova", Reggio Emilia
  - Ospedale Degli Infermi, Rimini
  - Fondazione PTV Policlinico Tor Vergata, Roma
  - AO San Camillo Forlanini, Roma
  - AOU S. Andrea Roma, Roma
  - Ospedale S. Eugenio, Roma
  - Policlinico Universitario Campus Bio-Medico, Roma
  - Roma Regina Elena IFO, Roma
  - Roma San Giovanni, Roma
  - Università degli Studi La Sapienza, Roma
  - Rozzano Humanitas, Rozzano
  - Siena, Siena
  - AOS Maria di Terni, Terni
  - AOS S. Giovanni Battista "Molinette", Torino
  - Azienda Ospedaliera Citta Della Salute E Della Scienza Di Torino, Torino
  - Ospedale Cardinale Panico, Tricase
  - Azienda Ospedaliera Univesritaria, Udine
  - Asst Settelaghi Ospedale Macchi, Varese
- Norway (2):
  - Oslo University Hospital, Oslo
  - St Olavs Hospital, Trondheim
- Warsaw Centrum Onkologi Instytucie, Warsaw, Poland
- Istituto Portugues de Oncologia de Lisboa, Lisbon, Portugal
- Lund Universitet, Lund, Sweden
- Switzerland (4):
  - IOSI, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Olten, Olten
  - Kantonsspital, Sankt Gallen
- Kyiv National Cancer Institute, Kiev, Ukraine
- United Kingdom (12):
  - Basingstoke & North Hamptshire Hospital, Basingstoke
  - Birmingham Heartlands Hospital, Birmingham
  - Glasgow Beatson Cancer Center, Glasgow
  - Leeds St. James's Hospital, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - Guy's & St. Thomas London, London
  - UCLH St. Thomas, London
  - Manchester The Christie NHS Foundation Trust, Manchester
  - Newcastle Freeman Hospital, Newcastle
  - Norfolk & Norwich University Hospital, Norfolk
  - Nottingham University Hospital, Nottingham
  - General Hospital, Southampton

REFERENCES:
- [Derived] Zucca E, Ceriani L, Ciccone G, Di Rocco A, Pirosa MC, Kriachok I, Botto B, Balzarotti M, Tucci A, Usai SV, Zilioli VR, Pennese E, Arcaini L, Dabrowska-Iwanicka A, Ferreri AJM, Merli F, Zhao W, Rigacci L, Cellini C, Hodgson D, Ionescu C, Minoia C, Lucchini E, Spina M, Fossa A, Janikova A, Cwynarski K, Mikhaeel NG, Jerkeman M, Stathis A, Cozens K, Ielmini N, De Martino I, Walewski J, Trneny M, Cavalli F, Ricardi U, Johnson PWM, Davies A, Martelli M. Impact of immunochemotherapy regimens on outcomes of patients with primary mediastinal B-cell lymphoma in the IELSG37 trial. Blood. 2025 Dec 4;146(23):2758-2764. doi: 10.1182/blood.2025028823. PMID 40939190
- [Derived] Martelli M, Ceriani L, Ciccone G, Ricardi U, Kriachok I, Botto B, Balzarotti M, Tucci A, Usai SV, Zilioli VR, Pennese E, Arcaini L, Dabrowska-Iwanicka A, Ferreri AJM, Merli F, Zhao W, Rigacci L, Cellini C, Hodgson D, Ionescu C, Minoia C, Lucchini E, Spina M, Fossa A, Janikova A, Cwynarski K, Mikhaeel G, Jerkeman M, Di Rocco A, Stepanishyna Y, Vitolo U, Santoro A, Re A, Puccini B, Olivieri J, Petrucci L, Barrington SF, Malkowski B, Metser U, Versari A, Chauvie S, Walewski J, Trneny M, Cavalli F, Gospodarowicz M, Johnson PWM, Davies A, Zucca E; International Extranodal Lymphoma Study Group (IELSG). Omission of Radiotherapy in Primary Mediastinal B-Cell Lymphoma: IELSG37 Trial Results. J Clin Oncol. 2024 Dec;42(34):4071-4083. doi: 10.1200/JCO-24-01373. Epub 2024 Aug 19. PMID 39159403